CLINICAL TRIAL: NCT03438487
Title: A Prospective Observational Safety Study on Pregnancy Outcomes in Women Immunized With Seasonal Cell Culture Influenza Trivalent (TIVc) or Quadrivalent (QIVc) Vaccine During Pregnancy
Brief Title: Flucelvax (TIVc or QIVc) Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Other Study IDs: V130_11OB
Record Dates: First submitted 2017-11-21; First posted 2018-02-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Influenza, Human; Pregnancy; Birth Defect
MeSH Terms: conditions — Influenza, Human; Congenital Abnormalities | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Flucelvax Trivalent or Quadrivalent Influenza Vaccine: Flucelvax Trivalent or Quadrivalent exposure in pregnancy
  Interventions: Biological: Flucelvax Trivalent Influenza Vaccine; Biological: Flucelvax Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Flucelvax Trivalent Influenza Vaccine — Flucelvax is a cell culture seasonal trivalent influenza vaccine that contains the following influenza hemagglutinin antigens: 1) A/H1N1-like virus, 2) A/(H3N2)-like virus, 3) B/Yamagata lineage or B/Victoria lineage
  Vaccine exposure in routine care (no vaccination per protocol)
  Other Names: Flucelvax
Biological: Flucelvax Quadrivalent Influenza Vaccine — Flucelvax Quadrivalent is a cell culture seasonal quadrivalent influenza vaccine that contains the following influenza hemagglutinin antigens: 1) A/H1N1-like virus, 2) A/(H3N2)-like virus, 3) B/Yamagata lineage, 4) B/Victoria lineage
  Vaccine exposure in routine care (no vaccination per protocol)
  Other Names: Flucelvax Quadrivalent

SUMMARY:
The study is a population based prospective cohort study designed to collect data on pregnancy outcomes and events of interest among women immunized with the TIVc or QIVc vaccine during pregnancy.

ELIGIBILITY:
Inclusion Criteria -

Enrollment and data collection will be coordinated through a coordination center (CC). The minimum eligibility criteria required for enrollment are as follows:

* Sufficient information to confirm that the exposure of interest occurred during pregnancy and at which date.
* Sufficient information to determine whether it concerns a prospectively enrolled subject, since retrospective cases are ineligible for enrollment.
* Reporter (e.g. HCP) contact information to allow for follow-up

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population will include pregnant women within the US who were immunized with the TIVc or the QIVc vaccine as part of routine care at any time during pregnancy. Eligible pregnant women may self-enroll or voluntarily be enrolled by their HCP.
  Women under 18 can be included in the study as long as parental consent can be obtained. De-identified data on minors will be accepted into the study if permitted by laws and regulations.
Sampling Method: Non-Probability Sample
Enrollment: 692 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Safety Objective: Number of cases for pregnancy outcomes among women immunized as part of routine care with the seasonal cell culture influenza trivalent (TIVc) or quadrivalent (QIVc) vaccine during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
  Number of cases for pregnancy outcomes will be reported as one of the following: live birth, stillbirth, spontaneous abortion and elective termination
Safety Objective: Number of cases with major congenital malformations among women immunized as part of routine care with the seasonal cell culture influenza trivalent (TIVc) or quadrivalent (QIVc) vaccine during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
Safety Objective: Number of cases with events of preterm birth among women immunized as part of routine care with the seasonal cell culture influenza trivalent (TIVc) or quadrivalent (QIVc) vaccine during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks
Safety Objective: Number of cases with low birth weight among women immunized as part of routine care with the seasonal cell culture influenza trivalent (TIVc) or quadrivalent (QIVc) vaccine during pregnancy. | From time of enrollment during pregnancy to time of delivery or pregnancy termination; a follow-up period of up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Head Epidemiology, Study Director — Seqirus
Locations (1):
- Syneos Health, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided